CLINICAL TRIAL: NCT05364138
Title: Evaluating Scaleup of an Adapted Breast Cancer Early Diagnosis Program in Rwanda
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners in Health (Other); Rwanda Biomedical Centre (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Lydia Pace, MD, MPH, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2021P002943
Record Dates: First submitted 2022-03-29; First posted 2022-05-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Benign Breast Disease; Cervix Cancer
Keywords: Rwanda; breast cancer; screening; early detection
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Breast cancer incidence is increasing in low- and middle-income countries (LMICs) and breast cancer mortality is high in these regions largely due to late stage diagnoses. This is true in the low-income East African country of Rwanda, where there are no national protocols in place to guide evaluation and referral of breast symptoms at primary health facilities.

This study will use quantitative and qualitative methods to examine implementation of the Women's Cancer Early Detection Program (WCEDP) in order to understand optimal strategies to scale and sustain breast cancer early diagnosis in Rwanda and other limited-resource settings. The WCEDP is an adaptation of a prior intervention in Burera District, which focused on building community awareness of breast symptoms, improving clinicians' clinical breast assessment (CBA) skills, and implementing weekly breast clinics at the primary health care center and hospital levels. The Burera intervention was associated with improvements in health care workers' knowledge and skills, increases in care-seeking and receipt of care by women with breast symptoms, and an increase in early-stage breast cancer diagnoses.

DETAILED DESCRIPTION:
Despite the Burera trial's promising results it was clear adaptations would be needed for real-world scaleup. The Burera intervention focused on breast health in isolation, hindering scalability in a limited-resource health system. In addition, it benefited from intensive patient tracking, feasible with the study's resources and implementation in a single district. Rwanda Biomedical Centre (RBC) is now scaling up breast cancer early diagnosis using the Burera training program with two key adaptations. First, in an effort to expand reach and increase efficiency, breast cancer early diagnosis services are offered together with cervical cancer screening in a combined initiative, the Women's Cancer Early Detection Program. The WCEDP combines these services through: 1)Combined provider trainings; 2)Community awareness-raising about both cancers; and 3)Weekly district hospital (DH) and HC clinics for women eligible for cervical cancer screening and CBA. RBC's second adaptation, an effort to facilitate patient tracking and linkage to care at scale, is a tablet-based EMR that allows clinicians to share information across facilities, identify missed visits, and document patient phone calls. These adaptations address priorities of the WHO's Global Breast Cancer Initiative: integrating early diagnosis into primary care services and building systems to facilitate referrals. By examining these adaptations in a real-world setting, this research will contribute to global efforts to identify evidence-based implementation strategies to address breast cancer in LMICs.

This study will leverage a longstanding partnership between RBC, Partners In Health (PIH), and Brigham and Women's Hospital (BWH) to pursue the following Specific Aims:

Aim 1. Use the RE-AIM framework to examine implementation and impact of Rwanda's adaptation and scale-up of breast cancer early diagnosis within the WCEDP, in 3 districts with 52 HCs.

1a. Evaluate the WCEDP's reach using interrupted time series analysis to examine its impact on the number of patients receiving CBA at HCs, and engagement of older women and those with breast symptoms.

1b. Examine program effectiveness, adoption and implementation by assessing timely linkage to care, loss-to-follow-up, service delivery, and EMR use.

Aim 2. Use patient and provider interviews, guided by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework, to elicit contextual factors related to successes and challenges of scaleup, including the WCEDP's fit and acceptability for communities, clinicians, and facilities.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who are evaluated for a breast concern or receive breast cancer screening through implementation of the nationally-led early detection programs

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is the population served by the health centers that are implementing the nationally-led breast cancer early detection program.
Sampling Method: Non-Probability Sample
Enrollment: 2357 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting to health centers for CBA per week (Reach) | 12 months
  The primary analysis will be interrupted time series (ITS) Poisson regression to compare the number of patients presenting for CBA to health centers each week in the months before and after initiation of the WCEDP

SECONDARY OUTCOMES:
Age of patients received (Reach) | 18 months
  The investigators will examine the median age of individuals presenting before and after WCEDP
Proportion of patients receiving CBA who had breast symptoms (Reach) | 18 months
  Investigators will examine the proportion of patients evaluated at health centers with CBA who had symptoms
Proportion of patients evaluated with CBA at health centers who also had cervical cancer screening (Reach) | 18 months
  Proportion of patients evaluated with CBA at health centers who also had cervical cancer screening (Reach)
WCEDP Effectiveness - HCs | 12 months
  Number and percentage of women seen at health centers for CBA who are referred to district hospitals (and seen within 1 month of DH visit)
WCEDP Effectiveness - DHs | 12 months
  Number and percentage of women seen at district hospitals for CBA who are referred to referral facilities (and seen within 1 month of DH visit)
WCEDP Adoption - CHWs | 12 months
  Number and percentage of community health workers (CHWs) trained
WCEDP Adoption - Clinicians | 12 months
  Number and percentage of clinicians trained in the program and in electronic medical record
WCEDP Implementation - Clinics | 6 and 12 months
  Number and percentage of weeks that clinics are held at each health center and district hospital (and the average percentage per district)
WCEDP Implementation - CHWs | 6 and 12 months
  Number of days/ month that CHWs hold community awareness events or do home visits (and average percentage per district)
WCEDP Implementation - electronic medical record | 6 and 12 months
  Proportion of weeks in which electronic medical record missed-visit reports are run in each district hospital
WCEDP Implementation - Phone calls | 6 and 12 months
  Of patients who have missed district hospital visits, percentage with phone call documented in the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Pace, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners in Health (Inshuti Mu Buzima), Butaro, Rwanda